CLINICAL TRIAL: NCT06396026
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TLL-018 in Participants With Moderate-to-Severe Chronic Spontaneous Urticaria With Inadequate Controll to Second Generation H1-antihistamines
Brief Title: A Study of Efficacy and Safety of TLL-018 in CSU Participants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLL-018-303
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Intervention Model Description: Drug: TLL-018 Drug: Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): TLL018 tablets,1piece,BID
  Interventions: Drug: TLL-018 tablets
- Arm 2 (Placebo Comparator): Placebo tablets,1piece,BID
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: TLL-018 tablets — Oral TLL-018 tablets taken orally 1 pieces BlD for 52 weeks
  Arms: Arm 1
Drug: Placebo tablets — Oral Placebo tablets taken orally 1 pieces BlD for 12 weeks and then Oral TLL-018 tablets taken orally 1 pieces BlD for 40 weeks.
  Arms: Arm 2

SUMMARY:
A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TLL-018 in Participants With Moderate-to-Severe Chronic Spontaneous Urticaria (CSU) With Inadequate Controll to Second Generation H1-antihistamines.

DETAILED DESCRIPTION:
This is a randomized, double-blind, single-dummy, placebo-parallel-group, phase 3 study to assess the safety and efficacy of TLL-018 in Moderate-to-Severe Chronic Spontaneous Urticaria (CSU) participants who had an Inadequate Controll to Second Generation H1-antihistamines.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75.
* Diagnosis of CSU refractory to secomd-generation H1-AH.
* CSU diagnosis for ≥ 6 months.
* The presence of itch and hivese despite current use of an approved dose of H1-AH prior to screening visit.
* UAS7 score (range 0-42) ≥ 16 and itch component of UAS7 (range 0-21) ≥ 8 during 7 days prior to randomization (Day 1).
* Participants were required to take a stable standard dose of a second generation H1-AH concomitantly according to local guidelines.
* Willing and able to complete UPDD for the duration of the study.
* Evidence of urticaria confirmed by the investigator prior to randomization.
* Women of Child Bearing Potential (WOCBP) should not be pregnant or breastfeeding and the pregnancy test should be negative before randomization.
* Participants (whether male or female) should have adequate barrier contraception during the whole treatment period and at least 90 days after treatment; subjects should avoid the sperm or ovum donation for at least six months after treatment.

Exclusion Criteria:

* Participants meeting Chinese Guidelines for Urticaria Diagnosis and Treatment with the following concomitant diseases cannot be enrolled:

  1. Clearly defined underlying etiology for chronic urticarias other than CSU. E.g. induced urticaria, including but not limited to artificial urticaria.
  2. Any disease, which may have symptoms of urticaria and/or angioedema, including but not limited to urticaria and vasculitis.
  3. Suffering from other chronic pruritic diseases that may affect the judgment of efficacy results, such as psoriasis, atopic dermatitis, etc.
  4. Previous malignancy, herpes zoster, active tuberculosis.
  5. Other symptoms of progressive or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, or cerebral disease.
  6. Taking part in this study, in the opinion of the investigator, places the patient at unacceptable risk.
* Participants with any of the following prior therapies or concomitant medications cannot be enrolled:

  1. Have received any study drug within 4 weeks or less than 5 elimination of half-life period before randomization (whichever is longer).
  2. Have received biological agent within 3 months or 5 elimination of half-life period prior to randomization (whichever is longer).
  3. Have received immunosuppressive/modulatory drug within 4 weeks before randomization.
  4. Have received any live vaccine within 2 months before randomization or plan to receive a live vaccine during the study.
* Have experienced major surgery within 4 weeks before randomization, or expected to receive major surgical treatment after enrollment;
* Have donated blood more than 400 ml or received blood transfusion within 3 months prior to the study.
* History of drug or alcohol abuse within 6 months prior to screening.
* Allergy to ingredients or excipients of H1-AH or TLL-018.
* Laboratory test results are abnormal and may interfere the study judged by investigators.
* Participants are not appropriate for participation in any other situation or condition in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in UAS7 at Week 12 | 12 weeks
  To demonstrate that TLL-018 is superior to placebo in CSU with respect to change from baseline in UAS7 at Week 12 by assessing absolute change from baseline in weekly Urticaria Activity Score (UAS7) at week 12.
  The UAS7 is a scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Change from baseline in ISS7 at Week 12 | 12 weeks
  To demonstrate that TLL-018 is superior to placebo in CSU with respect to change from baseline in ISS7 at Week 12 by assessing absolute change from baseline in weekly Itch Severity Score (ISS7) at week 12.
  The ISS7 is the itch severity score for 7 days, and it ranges from 0 to 21.

SECONDARY OUTCOMES:
Change from baseline in HSS7 at Week 12 | 12 weeks
  To demonstrate that TLL-018 is superior to placebo in CSU with respect to change from baseline in HSS7 at Week 12 by assessing absolute change from baseline in hive severity score (HSS7) at week 12.
  The HSS7 is the hive severity score for 7 days, and it ranges from 0 to 21.
Proportion of Participants With UAS7≤6 Response at Week 12 | 12 weeks
  To demonstrate that a greater proportion of participants achieve disease activity control UAS7≤6 at Week 12 who are treated with TLL-018 compared to placebo-treated participants by assessing achievement of UAS7≤6 at week 12.
Proportion of Participants With UAS7=0 Response at Week 12 | 12 weeks
  To demonstrate that a greater proportion of participants achieve complete absence of hives and itch (UAS7 = 0) at Week 12 who are treated with TLL-018 compared to placebo-treated participants by achievement of UAS7 = 0 at week 12.
Proportion of Participants With DLQI=0/1 Response at Week 12 | 12 weeks
  To demonstrate that a greater proportion of participants who are treated with TLL-018 achieve DLQI = 0/1 at Week 12 compared to placebo-treated participants by assessing achievement of DLQI = 0/1 at week 12.
Change from baseline in DLQI at Week 12 | 12 weeks
  To demonstrate that TLL-018 is superior to placebo in CSU with respect to change from baseline in DLQI at Week 12 by assessing absolute change from baseline in DLQI at week 12.
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | 52 weeks
  To demonstrate the safety and tolerability of TLL-018 by assessing occurrence of treatment emergent adverse events and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of Medical Sciences, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No